CLINICAL TRIAL: NCT06202456
Title: A Single-arm, Multicenter Phase IV Study to Investigate the Efficacy and Safety of Huazhi Rougan Granule in the Treatment of Non-alcoholic Simple Fatty Liver (Damp-heat Obstruction Syndrome: Shi-Re-Zhong-Zu Zheng)
Brief Title: A Phase IV Study of Huazhi Rougan Granule in the Treatment of Non-alcoholic Simple Fatty Liver
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-HZRG-G-IV
Record Dates: First submitted 2023-12-13; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Efficacy and Safety

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Huazhi Rougan granule (Experimental)
  Interventions: Drug: Huazhi Rougan granule

INTERVENTIONS:
Drug: Huazhi Rougan granule — Huazhi Rougan granule

SUMMARY:
An open Label, Single-arm, Multicenter phase IV study; There was a 2-week screening period and a 12-week / 24-week treatment period

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Those who meet the diagnostic criteria of non-alcoholic simple fatty liver and traditional chinese medicine syndrome classification of damp-heat obstruction syndrome;
3. Voluntarily sign informed consent;
4. Liver-to-spleen CT ratio < 1.0; The imaging findings of liver were consistent with the diagnostic criteria of diffuse fatty liver;
5. HbA1c≤6.5%；ALT、AST、TBil≤2×ULN；GFR≥60（ml/min/1.73m2）.

Exclusion Criteria:

1. Fatty liver caused by chronic heart failure, malnutrition and pregnancy, encephalopathy fatty liver syndrome (Reye syndrome), B-lipoprotein deficiency, localized fatty liver; Fatty liver caused by diabetes, long-term use of hormones, enteritis, gastrointestinal postoperative chronic infection, etc.; Small intestinal bypass surgery, hepatocyte toxicity injury, chronic febrile diseases such as tuberculosis, ulcerative nodules;
2. Severe fatty liver with ascites, edema, hyponatremia and other suspected cirrhosis; Hepatitis or cirrhosis caused by viruses, drug poisoning, immune diseases and other factors;
3. Pregnant and lactating women, women of childbearing age who do not take effective contraceptive measures (such as condoms, hormonal contraceptives, intrauterine devices) or male subjects who do not want to use contraception;；
4. Patient with serious primary cardiovascular disease, kidney disease and other serious diseases that affect survival;
5. Patient with a history of cancer;
6. Patient with HCV antibody, HIV antibody positive or HBsAg positive and HBV-DNA titer positive;
7. Have a history of alcohol abuse (alcohol equivalent male≥30g/d, female ≥20g/d) or drug abuse；
8. Allergic to the components of this drug；；
9. Those who participated in other clinical investigators within 3 months prior to screening;
10. Those who with a history of diabetes；
11. Patients who had used the same traditional Chinese medicine for the treatment of non-alcoholic simple fatty liver within 2 weeks before screening (except experimental drugs);
12. The investigators consider she/he inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2007 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Liver-to-spleen CT ratio | 12 weeks
  Clinical recovery: liver/spleen CT ratio ≥ 1; Obvious effect: liver/spleen CT ratio decreased by 2 grades (severe → mild); Effective: Liver/spleen CT ratio decreased by 1 grade (severe → moderate, or moderate → mild) :+ Ineffective: liver/spleen CT ratio did not change or even increased.

SECONDARY OUTCOMES:
The reduction of traditional Chinese medicine (TCM) syndrome integral | 12 weeks
  Clinical recovery: syndrome integral decreased ≥ 95%; Obvious Effective:70%≤the reduction of syndrome integral <95%; Effective :30%≤the reduction of syndrome score <70%; Ineffective: less than 30% reduction in syndrome integral. note: The reduction of TCM syndrome integral (%) = (Pre-treatment integral - post-treatment integral)/Pre-treatment integralx 100%
the reduction of ALT | 12 weeks
  Clinical control: Liver enzymology (ALT) returned to normal; + Obvious effect: liver enzyme (ALT) index decreased by ≥50%; Effective: Liver enzyme (ALT) index decreased <50% but≥ 30%; Ineffective: Liver enzyme (ALT) index decreased <30%。
the reduction of blood lipid index | 12 weeks
  blood lipid index including TC、TG、and HDL-C

CONTACTS AND LOCATIONS:
Locations (1):
- Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided